CLINICAL TRIAL: NCT06612879
Title: An Open-Label, Single Dose Study to Assess the Breast Milk and Plasma Pharmacokinetics of Omaveloxolone (BIIB141) in Healthy Lactating Women
Brief Title: A Study to Find Out How BIIB141 (Omaveloxolone) Moves From the Blood Into the Breastmilk of Healthy Women Who Are Breastfeeding or Pumping Milk
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 296HV101
Record Dates: First submitted 2024-09-23; First posted 2024-09-25 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — omaveloxolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Omaveloxolone (Experimental): Participants will receive a single oral dose of omaveloxolone on Day 1.
  Interventions: Drug: Omaveloxolone

INTERVENTIONS:
Drug: Omaveloxolone — Administered as specified in the treatment arm.
  Other Names: BIIB141; SKYCLARYS

SUMMARY:
In this study, researchers will learn how BIIB141, also known as omaveloxolone or SKYCLARYS®, moves through the body. This is a drug available for doctors to prescribe for patients with Friedrich's Ataxia. But, this drug has not yet been tested in women who have recently given birth and are breastfeeding or pumping milk for their babies. So, researchers do not know how much of the drug could be passed on to babies through the breastmilk of mothers who may take BIIB141.

The main objective of this study is to learn how a single dose of BIIB141 is processed in both the breastmilk and in the blood of healthy women who are breastfeeding.

The main question researchers want to answer in this study is:

* How does BIIB141 move from the blood into the breastmilk?

Researchers will also learn more about:

* How BIIB141 moves through the blood
* What dose of BIIB141 a baby may get from the mother's breastmilk
* Any medical problems the participants have during the study

This study will be done as follows:

* Participants will be screened to check if they can join the study. The screening period will be up to 28 days, after which participants will check into their study research center.
* Participants will take a single dose of BIIB141 as a tablet by mouth on Day 1.
* Participants will remain at their study research center for 6 days. During this time, the participants will be provided with an electric breast pump. This is so that the researchers can collect breastmilk samples before and after the participants take BIIB141. The researchers will also collect blood samples.
* After leaving the study research center, the participants will return every 2 days for the next 10 days for more tests and checkups.
* Finally, there will be a follow-up with a "lactation consultant" up to 30 days after each participant's last study visit. This is someone who can help participants with breastfeeding or pumping.
* Each participant will be in the study for up to 2.5 months.

ELIGIBILITY:
Key Inclusion Criteria:

* Lactating female 18 to 45 years of age.
* Has given birth to an infant of at least 37 weeks' gestation.
* Is at least 6 weeks postpartum by Day 1.
* Body mass index at screening between 18.0 and and < 35.0 kilograms per meter square (kg/m^2), inclusive.
* Is willing to discontinue breastfeeding their infant from check-in (Day -1) through 19 days after dosing.
* Has never taken omaveloxolone.

Key Exclusion Criteria:

* History of any clinically significant cardiovascular, endocrine, gastrointestinal, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, dermatologic, neurologic, psychiatric, or renal disease, or other major disease, as determined by the Investigator.
* Clinically significant (as determined by the Investigator) 12-lead electrocardiogram (ECG) abnormalities.
* History of, or positive test result at Screening for, human immunodeficiency virus.
* Chronic, recurrent, or serious infection (e.g., pneumonia, septicemia), as determined by the Investigator, within 90 days prior to Screening or between Screening and Day -1.
* Presence or history of hypotension or hypertension.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 12 (Actual)
Dates: Start 2024-10-18 (Actual); Primary Completion 2025-03-11 (Actual); Study Completion 2025-04-08 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Concentration (Cmax) of Omaveloxolone in Breast Milk | Predose and at multiple timepoints postdose (up to Day 15)
Time to Achieve Cmax (Tmax) of Omaveloxolone in Breast Milk | Predose and at multiple timepoints postdose (up to Day 15)
Average Concentration Based on Area Under the Concentration-Time Curve (AUC [Cav]) of Omaveloxolone in Breast Milk | Predose and at multiple timepoints postdose (up to Day 15)
Area Under the Concentration Time Curve From Time Zero to the Time of Last Measurable Concentration (AUC0-tlast) of Omaveloxolone in Breast Milk | Predose and at multiple timepoints postdose (up to Day 15)
Time of the Last Measurable Concentration (Tlast) of Omaveloxolone in Breast milk | Predose and at multiple timepoints postdose (up to Day 15)
AUC Time Curve From Time Zero to Infinity (AUCinf) of Omaveloxolone in Breast Milk | Predose and at multiple timepoints postdose (up to Day 15)
Milk-to-Plasma Ratio (M/P) of Omaveloxolone | Predose and at multiple timepoints postdose (up to Day 15)
Cumulative Amount of Omaveloxolone Excreted in Breast Milk (Ae) Over 24 Hours (Ae0-24) Postdose | At multiple timepoints postdose (up to 24 hours)
Cumulative Amount of Omaveloxolone Excreted in Breast Milk (Ae) Over 96 Hours (Ae0-96) Postdose | At multiple timepoints postdose (up to 96 hours)
Fraction of Omaveloxolone Excreted in Breast Milk (Fe) Over 24 Hours (Fe0-24) | At multiple timepoints postdose (up to 24 hours)
Fraction of Omaveloxolone Excreted in Breast Milk (Fe) Over 96 Hours (Fe0-96) | At multiple timepoints postdose (up to 96 hours)

SECONDARY OUTCOMES:
Cmax of Omaveloxolone in Plasma | Predose and at multiple timepoints postdose (up to Day 15)
Tmax of Omaveloxolone in Plasma | Predose and at multiple timepoints postdose (up to Day 15)
AUC[Cav] of Omaveloxolone in Plasma | Predose and at multiple timepoints postdose (up to Day 15)
AUC0-tlast of Omaveloxolone in Plasma | Predose and at multiple timepoints postdose (up to Day 15)
AUCinf of Omaveloxolone in Plasma | Predose and at multiple timepoints postdose (up to Day 15)
Terminal Elimination Rate Constant (λz) of Omaveloxolone in Plasma | Predose and at multiple timepoints postdose (up to Day 15)
Apparent Plasma Terminal Elimination Half-Life (t1/2) of Omaveloxolone | Predose and at multiple timepoints postdose (up to Day 15)
Apparent Plasma Clearance After Extravascular Administration (CL/F) of Omaveloxolone | Predose and at multiple timepoints postdose (up to Day 15)
Apparent Volume of Distribution During the Terminal Elimination Phase After Extravascular Administration (Vz/F) of Omaveloxolone | Predose and at multiple timepoints postdose (up to Day 15)
Percent of Area Under the Plasma Concentration-Time Curve From Time Zero Extrapolated to Infinity (AUC%extrap) of Omaveloxolone | Predose and at multiple timepoints postdose (up to Day 15)
Plasma Unbound Fraction (fu,p) of Omaveloxolone | Predose and at multiple timepoints postdose (up to Day 15)
Cmax of Unbound Plasma Fraction (Cmax,u) of Omaveloxolone | Predose and at multiple timepoints postdose (up to Day 15)
Cav of Unbound Plasma Fraction (AUCinf,u) of Omaveloxolone | Predose and at multiple timepoints postdose (up to Day 15)
AUC0-tlast of Unbound Plasma Fraction (AUC0-last,u) of Omaveloxolone in Plasma | Predose and at multiple timepoints postdose (up to Day 15)
AUCinf of Unbound Plasma Fraction (AUCinf,u) of Omaveloxolone | Predose and at multiple timepoints postdose (up to Day 15)
Estimated Daily Infant Dosage (DID) of Omaveloxolone | Predose and at multiple timepoints postdose (up to Day 15)
Relative Infant Dose (RID) of Omaveloxolone | Predose and at multiple timepoints postdose (up to Day 15)
Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | From Day 1 up to end of study follow-up (up to 45 days)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (1):
- Fortrea Madison WI, CRU, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/